CLINICAL TRIAL: NCT04038307
Title: Pre-emptive Intravenous Paracetamol for Prevention of Intraoperative Shoulder Tip Pain in Patients Undergoing Caesarean Section: A Randomized Double Blind Controlled Clinical Trial.
Brief Title: Pre-emptive Paracetamol for Prevention of Intraoperative Shoulder Tip Pain
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmin Hassab elnaby, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MS-12-2019
Record Dates: First submitted 2019-07-24; First posted 2019-07-30 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Cesarean Section
Keywords: shoulder tip pain
MeSH Terms: interventions — Acetaminophen; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Placebo Comparator): will receive 100 ml of saline
  Interventions: Drug: Saline Solution
- paracetamol group (Experimental): will receive 1gm paracetamol (100ml)
  Interventions: Drug: paracetamol

INTERVENTIONS:
Drug: paracetamol — 1gm
  Arms: paracetamol group
Drug: Saline Solution — 100ml
  Arms: control

SUMMARY:
the aim is to determine the efficacy of Paracetamol in reducing the incidence and severity of intraoperative shoulder pain in patients undergoing cesarean section.

DETAILED DESCRIPTION:
pregnant females scheduled for cesarean section under spinal anesthesia will be enrolled . two groups of patents will be recruited . the study group will receive paracetamol pre operative .

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women (ASA II) having singleton pregnancy at term (≤ 37 weeks of gestation) aged between 18 and 40 years.

Exclusion Criteria:

* Patients having allergy to study drug,
* gestational diabetes
* cardiovascular or biliary disorders
* asthma
* renal impairment
* preeclampsia
* any chronic pain condition or trauma in the shoulder, forearms or upper limbs
* patients with any contraindication to SA were excluded from the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
incidence shoulder tip pain | intraoperative
  presence of shoulder tip pain

SECONDARY OUTCOMES:
numerical rating scale | intraoperative
  severity of shoulder tip pain (0-10) where 0 is no pain and 10 is the worst pain ever

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No